CLINICAL TRIAL: NCT01745822
Title: Phase 3, Randomized Clinical Trial to Assess the Efficacy and Safety of Tenofovir in Hepatitis B Virus Infected, s and e Antigen Positive, Pregnant Women to Prevent Perinatal Transmission Despite Infant Passive-active HBV Immunization.
Brief Title: Maternal Antiviral Prophylaxis to Prevent Perinatal Transmission of Hepatitis B Virus in Thailand
Acronym: iTAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Chargé de recherches, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01HD071889 (NIH); U01HD071889 (NIH)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis B Chronic Infection; Pregnancy
Keywords: Hepatitis B; Hepatitis B sAg; Hepatitis B eAg; pregnancy
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir disoproxil fumarate (Experimental): tenofovir disoproxil fumarate, 300 mg tablets
  Interventions: Drug: tenofovir disoproxil fumarate
- Placebo (Placebo Comparator): matching placebo (of tenofovir disoproxil fumarate)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate — administration: tablet 300 mg, once a day, from enrollment at 28 weeks' gestation until 2 months postpartum
  Other Names: Viread; TDF; tenofovir
  Arms: Tenofovir disoproxil fumarate
Drug: placebo — administration: one tablet, once a day, from enrollment at 28 weeks' gestation until 2 months postpartum
  Arms: Placebo

SUMMARY:
Chronic hepatitis B (CHB) infection is complicated by cirrhosis and liver cancer. In Thailand, 7% of adults are chronically infected by Hepatitis B virus (HBV). The risk of perinatal transmission of HBV is about 12% when a mother has a high HBV load in her plasma, even if her infant receive specific immunoglobulin and vaccine.

The hypothesis of this study is that a potent antiviral, tenofovir, can decrease HBV load in HBV infected pregnant women and therefore reduce the risk of perinatal transmission/ Pregnant women participating in this study will receive tenofovir or placebo during the last trimester of pregnancy and two months postpartum. The risk of perinatal transmission will be compared between the two groups.

The results of the study will help define policy to manage HBV infected pregnant women to prevent perinatal transmission.

DETAILED DESCRIPTION:
This is a phase III, placebo controlled, double blind, randomized clinical trial to assess the efficacy and safety of tenofovir disoproxil fumarate (TDF) given from 28 weeks' gestation until 2 months postpartum to pregnant women with Hepatitis B (HB) virus (HBV) chronic infection and positive for HB s and e antigen to prevent perinatal transmission of HBV to their infants. All infants will receive HBV passive (HB specific immunoglobulin) and active (vaccine) immunization.

Chronic hepatitis B (CHB) infection is complicated by cirrhosis and hepatocellular carcinoma (HCC), the 10th leading cause of death worldwide.

In 2011, about 7% of adults in Thailand were HBsAg carriers. Infant hepatitis B (HB) immunization and HB immune globulin (HBIg) administered at birth effectively prevent most mother-to-child transmission (MTCT) of HBV. However, about 12% of mothers with high load of HBV transmit the virus to their infants, despite active and passive immunization.

Studies have suggested that antiviral treatment at the end of pregnancy and during early postpartum can reduce the risk of transmission to the child. A potential limitation to this approach is the risk of hepatic disease exacerbation following discontinuation of antiviral treatment postpartum, and this risk has not been properly evaluated. No randomized clinical trials have adequately demonstrated the efficacy and safety of maternal antiviral treatment the prevention of mother to child transmission of HBV. This is the reason why this approach is not currently recommended by the Associations for the Study of Liver Diseases.

We hypothesize that a potent antiviral, tenofovir, can decrease HBV viral load in HBV infected pregnant women and therefore reduce the risk of perinatal transmission, before infants are definitely protected by passive-active immunization. We also hypothesize that only moderate exacerbations of liver disease will be observed after discontinuation of a short antiviral course (5 months). While the primary objective of the study is to assess the efficacy of tenofovir versus placebo for the prevention of perinatal transmission, an important secondary objective is the assessment of the risk of postpartum hepatic disease exacerbation.

Within 2 years, 328 women and their infants will be enrolled from public hospitals in Thailand and randomized to receive either tenofovir disoproxil fumarate or matching placebo from 28 weeks of pregnancy until 2 months postpartum. Mothers and infants will be followed until one year postpartum.

The primary endpoint will be the detection of HBsAg and HBV DNA in infants at six months of life. An interim analysis will be conducted when half of the outcomes are available.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* At least 18 years of age
* Negative Human Immunodeficiency Virus (HIV) serology
* Positive HBsAg and hepatitis B e antigen (HBeAg) tests
* Gestational age of 28 weeks (+ or - 10 days) as determined by obstetrician
* Alanine Aminotransferase (ALT)≤30 U/L, confirmed ≤60 U/L on a subsequent blood draw
* Agreeing to bring their infants at the planned study visits at one study site until one year after delivery and to inform the site investigators if they plan to move to another place and not be able to return to the clinic.
* Understanding the need for adequate infant immunization and agreeing to the blood draws from their infants and the need for close follow up to manage possible exacerbation of hepatitis.

Exclusion Criteria:

* History of tenofovir treatment at any time, or any other anti-HBV treatment during the current pregnancy
* Creatinine clearance <50 ml/min, calculated using the Cockcroft-Gault formula
* Dipstick proteinuria>1+ (>30 mg/dL) or normoglycemic glucosuria confirmed on two separate occasions
* Positive serology for Hepatitis C infection less than 12 months prior to enrollment
* Evidence of pre-existing fetal anomalies incompatible with life
* Any concomitant condition or treatment that, in the view of the clinical site investigator, would contraindicate participation or satisfactory follow up in the study.
* Concurrent participation in any other clinical trial without written agreement of the two study teams

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague Jourdain, MD, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (17):
- Thailand (17):
  - Banglamung Hospital, Bang Lamung, Changwat Chon Buri
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Mae Chan Hospital, Mae Chan, Chiangrai
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima, Nakhon Ratchasrima
  - Bhumibol Adulyadej Hospital, Bangkok
  - Nopparat Rajathanee Hospital, Bangkok
  - Prapokklao Hospital, Chanthaburi
  - Health Promotion Center Region 10, Chiang Mai
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Chonburi Regional Hospital, Chon Buri
  - Khon Kaen Hospital, Khon Kaen
  - Lampang Hospital, Lampang
  - Lamphun Hospital, Lamphun
  - Samutprakarn Hospital, Mueang Samut Prakan
  - Phayao Provincial Hospital, Phayao
  - Samutsakhon Hospital, Samut Sakhon

IPD SHARING:
Plan to Share IPD: Undecided
Pending completion of analysis planned in the protocol

REFERENCES:
- [Background] Jourdain G, Ngo-Giang-Huong N, Cressey TR, Hua L, Harrison L, Tierney C, Salvadori N, Decker L, Traisathit P, Sirirungsi W, Khamduang W, Bowonwatanuwong C, Puthanakit T, Siberry GK, Watts DH, Murphy TV, Achalapong J, Hongsiriwon S, Klinbuayaem V, Thongsawat S, Chung RT, Pol S, Chotivanich N. Prevention of mother-to-child transmission of hepatitis B virus: a phase III, placebo-controlled, double-blind, randomized clinical trial to assess the efficacy and safety of a short course of tenofovir disoproxil fumarate in women with hepatitis B virus e-antigen. BMC Infect Dis. 2016 Aug 9;16:393. doi: 10.1186/s12879-016-1734-5. PMID 27506549
- [Result] Jourdain G, Ngo-Giang-Huong N, Harrison L, Decker L, Tierney C, Cressey TR, Achalapong J, Siberry GK, Nelson NP, and Chotivanich N. TDF to prevent perinatal hepatitis B virus transmission: a randomized trial (iTAP). Conference on Retroviruses and Opportunistic Infections (CROI) Abstract 584LB; 2017 February 13; Seattle, WA, USA. http://www.croiconference.org/sessions/tdf-prevent-perinatal-hepatitis-b-virus-transmission-randomized-trial-itap
- [Result] Jourdain G, Ngo-Giang-Huong N, Harrison L, Decker L, Khamduang W, Tierney C, Salvadori N, Cressey TR, Sirirungsi W, Achalapong J, Yuthavisuthi P, Kanjanavikai P, Na Ayudhaya OP, Siriwachirachai T, Prommas S, Sabsanong P, Limtrakul A, Varadisai S, Putiyanun C, Suriyachai P, Liampongsabuddhi P, Sangsawang S, Matanasarawut W, Buranabanjasatean S, Puernngooluerm P, Bowonwatanuwong C, Puthanakit T, Klinbuayaem V, Thongsawat S, Thanprasertsuk S, Siberry GK, Watts DH, Chakhtoura N, Murphy TV, Nelson NP, Chung RT, Pol S, Chotivanich N. Tenofovir versus Placebo to Prevent Perinatal Transmission of Hepatitis B. N Engl J Med. 2018 Mar 8;378(10):911-923. doi: 10.1056/NEJMoa1708131. PMID 29514030
- [Result] Jourdain G, Harrison LJ, Ngo-Giang-Huong N, Cressey TR, Decker L, Tierney C, Achalapong J, Kanjanavikai P, Luvira A, Srirompotong U, Murphy TV, Nelson N, Siberry GK, Pol S, for the iTAP Study Group. iTAP trial: maternal and infant efficacy and safety results 12 months after delivery. CROI, 4-7 March 2018, Boston, USA. #1316, Oral Presentation O-11
- [Result] Salvadori N, Fan B, Teeyasoontranon W, Ngo-Giang-Huong N, Phanomcheong S, Luvira A, Puangsombat A, Suwannarat A, Srirompotong U, Putiyanun C, Kourtis A, Bulterys M, Siberry GK, Jourdain G. TDF prophylaxis for PMTCT of HBV: effect on maternal and infant bone mineral density. CROI, 4-7 March 2018, Boston, USA. #1174. Poster and Themed Discussion TD-09
- [Result] Cressey TR, Harrison L, Achalapong J, Kanjanavikai P, Patamasingh Na Ayudhaya O, Liampongsabuddhi P, Siriwachirachai T, Putiyanun C, Suriyachai P, Tierney C, Salvadori N, Chinwong D, Decker L, Tawon Y, Murphy TV, Ngo-Giang-Huong N, Siberry GK, Jourdain G; iTAP Study Team. Tenofovir Exposure during Pregnancy and Postpartum in Women Receiving Tenofovir Disoproxil Fumarate for the Prevention of Mother-to-Child Transmission of Hepatitis B Virus. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01686-18. doi: 10.1128/AAC.01686-18. Print 2018 Dec. PMID 30275094
- [Result] Salvadori N, Fan B, Teeyasoontranon W, Ngo-Giang-Huong N, Phanomcheong S, Luvira A, Puangsombat A, Suwannarat A, Srirompotong U, Putiyanun C, Cressey TR, Decker L, Khamduang W, Harrison L, Tierney C, Shepherd JA, Kourtis AP, Bulterys M, Siberry GK, Jourdain G. Maternal and Infant Bone Mineral Density 1 Year After Delivery in a Randomized, Controlled Trial of Maternal Tenofovir Disoproxil Fumarate to Prevent Mother-to-child Transmission of Hepatitis B Virus. Clin Infect Dis. 2019 Jun 18;69(1):144-146. doi: 10.1093/cid/ciy982. PMID 30924492
- [Result] Ngo-Giang-Huong N, Salvadori N, Khamduang W, Cressey TR, Harrison LJ, Decker L, Tierney C, Jullapong A, Murphy TV, Nelson N, Siberry GK, Chung RT, Pol S, Jourdain G. Hepatitis B virus DNA level changes in HBeAg+ pregnant women receiving TDF for PMTCT. Conference on Retroviruses and Opportunistic Infections (CROI), Seattle, WA, 4-7 Mar 2019
- [Result] Bukkems V, Smolders E, Jourdain G, Hawkins D, Achalapong J, Kanjanavikai P, Taylor G, Prommas S, Burger D, Colbers A, Cressey TR, for the iTAP Study Team & PANNA network. Tenofovir plasma concentrations in pregnant women: comparison of hepatitis B and HIV-infected patients. 20th International Workshop on Clinical Pharmacology of HIV, Hepatitis & Other Antiviral Drugs. Noordwijk, the Netherlands, 14-16-May 2019
- [Result] Jourdain G, Traisathit P, Salvadori N, Wangsaeng N, Khamduang W, Ngo-Giang-Huong N, for the iTAP Study Group. Immunization response in infants born to HBsAg+ and HBeAg+ mothers receiving TDF (ID 3681). Conference on Retroviruses and Opportunistic Infections (CROI), Hynes Convention Center, USA, 8-11 Mar 2020, Virtual Conference
- Available data/document: Individual Participant Data Set — https://dash.nichd.nih.gov/study/17511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Enrollment Dates: January 8, 2013 to August 19, 2015 in 17 hospital based antenatal care and pediatrics departments in Thailand
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Started | 331 (168 mothers and 163 infants) | 323 (163 mothers and 160 infants)
Completed | 331 | 323
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Mothers only
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo | Total
Number analyzed (Participants) | 168 | 163 | 331
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.5 [22.6 to 29.1] | 26.7 [23.5 to 30.5] | 26.1 [22.9 to 30.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 163 | 331
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 168 | 163 | 331
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 28.3 [27.9 to 28.6] | 28.1 [27.9 to 28.6] | 28.3 [27.9 to 28.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With Hepatitis B Infection at 6 Months of Age
Description: Infection is defined as a HBsAg positive test confirmed by detectable HBV DNA
Time Frame: 6 months of age
Population: Participants in the primary analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 147 | 147
Participants | 0 | 3

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Occurrence of maternal and infant adverse events, including maternal and infants Serious Adverse Events (as defined by the International Conference on Harmonization Good Clinical Practice) and NIH Division of AIDS grade 3/4 signs and symptoms, regardless of their relatedness to the study treatment.
Time Frame: from enrollment (28 weeks' gestation) to 12 months postpartum
Population: Mother-infant pairs
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 329 | 323
Participants
  Maternal: number analyzed (Participants) | 168 | 163
  Maternal | 41 | 44
  Infant: number analyzed (Participants) | 161 | 160
  Infant | 43 | 38

3. Secondary Outcome: Percentage of Participants With Flares After Study Treatment Interruption
Description: Flare, or acute exacerbation of hepatitis B, after study treatment interruption is defined as an Alanine Aminotransferase plasma level above 300 IU/mL
Time Frame: Following planned discontinuation of study treatment up to 12 months postpartum
Population: Women who had delivered
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 154 | 157
Participants | 9 | 5

4. Secondary Outcome: Percentage of Infants With Hepatitis B Infection at or After 6 Months Through 12 Months of Age
Description: Infants will be considered HBV infected if at any time point at or after 6 months through 12 months of age, a sample tests positive for HBsAg and HBV DNA
Time Frame: at or after 6 months through 12 months of age
Population: infants until 12 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 147 | 147
Participants | 0 | 3

5. Secondary Outcome: Weight, Height and Head Circumference for Age
Description: Weight, length/height and head circumference WHO Z scores are measures of relative weight, height and head circumference adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: assessed at 6 months and 12 months of age, 6 months reported
Population: infants at 6 months of age
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
Number analyzed (Participants) | 148 | 146
Z-score
  Weight for age | -0.4 (1.1) | -0.2 (1.1)
  Length for age | -0.2 (1.2) | -0.2 (1.2)
  Head circumference for age | -0.6 (1.1) | -0.6 (0.9)

ADVERSE EVENTS:
Time Frame: From enrollment (28 weeks' gestation) to 12 months postpartum
Description: Adverse event information was collected using the same definitions of adverse event and serious adverse event as the clinicaltrials.gov definitions. Only serious adverse events and other (not including serious) Grade 3 or 4 adverse events are reported.
Arm/Group | Tenofovir Disoproxil Fumarate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/331 | 0/323
Serious Adverse Events (participants affected / at risk) | 62/331 | 66/323
Other Adverse Events (participants affected / at risk) | 42/331 | 31/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate (N=331) | Placebo (N=323)
Leukocytosis (Blood and lymphatic system disorders) | 2 | 4
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 4 | 1
Hemivertebra (Congenital, familial and genetic disorders) | 0 | 1
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 1 | 1
Talipes (Congenital, familial and genetic disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 1
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 4 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Endometritis decidual (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 0
Omphalitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4
Pneumonia viral (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 8 | 9
Treponema test positive (Investigations) | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 17 | 15
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 | 7
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Uterine inflammation (Reproductive system and breast disorders) | 0 | 1
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate (N=331) | Placebo (N=323)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Persistent foetal circulation (Congenital, familial and genetic disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 24 | 16
Aspartate aminotransferase increased (Investigations) | 3 | 3
Blood phosphorus decreased (Investigations) | 1 | 2
Neutrophil count abnormal (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT01745822/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT01745822/SAP_001.pdf